CLINICAL TRIAL: NCT04195464
Title: Effects of Dry Needling on Muscle Function in Patients With Hip Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Zaragoza (Other)
Responsible Party: Principal Investigator, Luis Ceballos Laita, Ph.D, Universidad de Zaragoza
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Universidad de Valladolid
Record Dates: First submitted 2019-12-04; First posted 2019-12-11 (Actual); Last update posted 2020-05-13 (Actual); Status verified 2020-05

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis | interventions — Dry Needling

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Doble-blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- DN (Experimental)
  Interventions: Other: Dry needling
- Sham-DN (Sham Comparator)
  Interventions: Other: Sham dry needling
- Control (No Intervention)

INTERVENTIONS:
Other: Dry needling — Dry needling is a skilled intervention that uses a thin filiform needle to penetrate the skin and stimulate underlying myofascial trigger points, muscular, and connective tissues for the management of neuromusculoskeletal pain and movement impairments
  Arms: DN
Other: Sham dry needling — Sham Dry needling use a non-penetrating acupuncture needle
  Arms: Sham-DN

SUMMARY:
The aim of this study was to assess the effects of dry needling technique on muscle strength and muscle length in patients with hip osteoarthritis at short term.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed medically with a X-Ray test
* American College of Rheumatology Criteria

Exclusion Criteria:

* Secondary osteoarthritis by a traumatism, Paget disease, inflammatory or metabolic disease, congenital diseases etc.
* Vascular or neurological disease.
* Musculoskeletal pathologies in lumbar spine, pelvis or lower limbs
* Fear of needles

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2019-12-11 (Actual); Primary Completion 2020-01-14 (Actual); Study Completion 2020-02-10 (Actual)

PRIMARY OUTCOMES:
muscle strength | Baseline
  The examiners assess the muscle strength using a hand-held dynamometer (model 01165) for hip internal and external rotation, flexion, extension, abduction and adduction.
muscle strength | up to 3 weeks
  The examiners assess the muscle strength using a hand-held dynamometer (model 01165) for hip internal and external rotation, flexion, extension, abduction and adduction.
Physical function | Baseline
  the examiners assess the physical function using the TImed Up and Go (TUG test) and the 40 meters-self-placed test .
Physical function | up to 3 weeks
  the examiners assess the physical function using the TImed Up and Go (TUG test) and the 40 meters-self-placed test .
Pain intensity | Baseline
  The examiners assess pain intensity after physical function tests using visual analogue scale
Pain intensity | up to 3 weeks
  The examiners assess pain intensity after physical function tests using visual analogue scale
Functional capacity with a validated questionnaire (WOMAC) | Baseline
  The examiners assess pain, stifness and functional capacity using the Western Ontario y McMaster Questionnaire
Functional capacity with a validated questionnaire (WOMAC) | Up to 3 weeks
  The examiners assess pain, stifness and functional capacity using the Western Ontario y McMaster Questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Luis Ceballos Laita, Soria, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ceballos-Laita L, Jimenez-Del-Barrio S, Marin-Zurdo J, Moreno-Calvo A, Marin-Bone J, Albarova-Corral MI, Estebanez-de-Miguel E. Effectiveness of Dry Needling Therapy on Pain, Hip Muscle Strength, and Physical Function in Patients With Hip Osteoarthritis: A Randomized Controlled Trial. Arch Phys Med Rehabil. 2021 May;102(5):959-966. doi: 10.1016/j.apmr.2021.01.077. Epub 2021 Feb 7. PMID 33567336